CLINICAL TRIAL: NCT04872569
Title: Pilot Testing A Pregnancy Decision Making Tool for Women With Spinal Cord Injury
Brief Title: Pilot Testing A Pregnancy Decision Making Tool for Women With Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Claire Z. Kalpakjian, Associate Chair, Department of Physical Medicine and Rehabilitation and Associate Professor of Physical Medicine and Rehabilitation, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00194755
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injuries; Pregnancy Related
Keywords: Decision tool
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision-making tool (Experimental): Women will receive the decision making tool and use for a 3 month period.
  Interventions: Behavioral: Decision-making tool

INTERVENTIONS:
Behavioral: Decision-making tool — Participants will be directed to use the decision tool for 3 months using it at their own pace.
  The tool covers topics relevant to women with disabilities in considering or planning a pregnancy and reflects core elements of decision making tools based on the Ottawa Framework for Decision Support.

SUMMARY:
The purpose of this project is to pilot test a decision-making tool that is tailored for women with SCI to support them in the decision-making process. Pilot testing focuses on feasibility and preliminary efficacy.

DETAILED DESCRIPTION:
The purpose of this project is to pilot test a decision-making tool that is tailored for women with SCI to support them in the decision-making process. Pilot testing focuses on feasibility and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury (traumatic or non-traumatic)
* Need for assistance with daily life activities and/or personal care; women with mild, moderate or severe severity will be eligible
* actively planning or in the process of making a decision about whether or not to get pregnant in the near future

Exclusion Criteria:

- No plans for getting pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Kalpakjian, PhD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Decision-making Tool: Women will receive the decision making tool and use for a 3 month period.
  Decision-making tool: Participants will be directed to use the decision tool for 3 months using it at their own pace.
  The tool covers topics relevant to women with SCI considering or planning a pregnancy and reflects core elements of decision making tools based on the Ottawa Framework for Decision Support.
Period: Overall Study
Arm/Group | Decision-making Tool
Started | 23
Completed | 21
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Decision-making Tool: Women will receive the decision making tool and use for a 3 month period.
  Decision-making tool: Participants will be directed to use the decision tool for 3 months using it at their own pace.
  The tool covers topics relevant to women with SCI in considering or planning a pregnancy and reflects core elements of decision making tools based on the Ottawa Framework for Decision Support.
Arm/Group | Decision-making Tool
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Count by sex: Female | 23
  Count by sex: Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23
Decisional Conflict Scale, Values Clarity sub-scale [Mean (Standard Deviation); unit: units on a scale] — The Decisional Conflict Scale is a self-report measure. Decisional conflict refers to a state of uncertainty about a course of action. For this study, this refers to uncertainty about pursuing a future pregnancy. The Values Clarity sub-scale refers to how much a respondent is clear about the values that guide their decision-making. Sub-scale items (3) are rated on 5-point Likert scales (ranging from strongly agree [5] to strongly disagree [1]) and summed for a total score range of 3 to 15. Higher scores represent greater clarity of values.
  units on a scale | 12.9 (1.7)
Decisional Conflict Scale, Support for Decision Making sub-scale [Mean (Standard Deviation); unit: units on a scale] — The Decisional Conflict Scale is a self-report measure. Decisional conflict refers to a state of uncertainty about a course of action. For this study, this refers to uncertainty about pursuing a future pregnancy. The Support for Decision Making sub-scale refers to how much support a respondent has from others about their decision-making. Sub-scale items (3) are rated on 5-point Likert scales (ranging from strongly agree [5] to strongly disagree [1]) and summed for a total score range of 3 to 15. Higher scores represent greater support for decision-making.
  units on a scale | 12.1 (2.3)
Decisional Conflict Scale, Uncertainty about the Decision sub-scale [Mean (Standard Deviation); unit: units on a scale] — The Decisional Conflict Scale is a self-report measure. Decisional conflict refers to a state of uncertainty about a course of action. For this study, this refers to uncertainty about pursuing a future pregnancy. The Uncertainty about the decision sub-scale refers to how much a respondent is uncertain about the decision. Sub-scale items (3) are rated on 5-point Likert scales (ranging from strongly agree [5] to strongly disagree [1]) and summed for a total score range of 3 to 15. Higher scores represent greater certainty about the decision.
  units on a scale | 9.9 (3.7)
Stage of Decision-Making Scale [Mean (Standard Deviation); unit: units on a scale] — The Stage of Decision Making is a single item self-report measure. The options range from "haven't begun to think about choices" to "have already made a decision and unlikely to change my mind". The instructions were modified to refer to pregnancy and excluded the first two options of not having begun to think about choices given inclusion criteria. For this study, the scale ranged from 1 (are considering the decision now) to 4 (have already made a decision and am unlikely to change my mind). A higher score reflects greater readiness to make a decision.
  units on a scale | 2.6 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Final Decisional Conflict Scale Score - Values Clarity Sub-scale
Description: The Decisional Conflict Scale is a self-report measure. Decisional conflict refers to a state of uncertainty about a course of action. For this study, this refers to uncertainty about pursuing a future pregnancy. The Values Clarity sub-scale refers to how much a respondent is clear about the values that guide their decision-making. Sub-scale items (3) are rated on 5-point Likert scales (ranging from strongly agree [5] to strongly disagree [1]) and summed for a total score range of 3 to 15. Higher scores represent greater clarity of values.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Women Using Tool: Women using the tool
Arm/Group | Women Using Tool
Number analyzed (Participants) | 21
units on a scale | 13.4 (1.6)

2. Primary Outcome: Final Decisional Conflict Scale Score - Support Sub-scale
Description: The Decisional Conflict Scale is a self-report measure. Decisional conflict refers to a state of uncertainty about a course of action. For this study, this refers to uncertainty about pursuing a future pregnancy. The Support for Decision Making sub-scale refers to how much support a respondent has from others about their decision-making. Sub-scale items (3) are rated on 5-point Likert scales (ranging from strongly agree [5] to strongly disagree [1]) and summed for a total score range of 3 to 15. Higher scores represent greater support for decision-making.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Decision Making Tool: Women using the tool for 12 weeks.
Arm/Group | Decision Making Tool
Number analyzed (Participants) | 21
units on a scale | 13.1 (2.0)

3. Primary Outcome: Final Decisional Conflict Scale Score - Uncertainty Sub-scale
Description: The Decisional Conflict Scale is a self-report measure. Decisional conflict refers to a state of uncertainty about a course of action. For this study, this refers to uncertainty about pursuing a future pregnancy. The Uncertainty about the decision sub-scale refers to how much a respondent is uncertain about the decision. Sub-scale items (3) are rated on 5-point Likert scales (ranging from strongly agree [5] to strongly disagree [1]) and summed for a total score range of 3 to 15. Higher scores represent greater certainty about the decision.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Making Tool
Number analyzed (Participants) | 21
units on a scale | 11.8 (3.3)

4. Primary Outcome: Final Readiness to Make a Choice in Stage of Decision-Making Scale
Description: The Stage of Decision Making is a single item self-report measure. The options range from "haven't begun to think about choices" to "have already made a decision and unlikely to change my mind". The instructions were modified to refer to pregnancy and excluded the first two options of not having begun to think about choices given inclusion criteria. For this study, the scale ranged from 1 (are considering the decision now) to 4 (have already made a decision and am unlikely to change my mind). A higher score reflects greater readiness to make a decision.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Making Tool
Number analyzed (Participants) | 21
units on a scale | 3.19 (1.1)

5. Secondary Outcome: Feasibility - Acceptability
Description: Acceptability of decision making tool is refers to whether the intervention is agreeable or satisfactory. In this study we measured this by self-report. We used 13 items that measured the presentation of information of the tool rated on Likert scales ranging from 1 (poor) to 4 (excellent) which are summed across all items. Possible scores can range from 13 to 52, with higher scores reflecting better information presentation.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Making Tool
Number analyzed (Participants) | 21
units on a scale | 38.96 (6.5)

6. Secondary Outcome: Feasibility - Demand
Description: Demand refers to the likelihood of using an intervention after the study is over. For this study, it is a single item rated on Likert scales of 1 (definitely not likely) to 5 (very likely). Higher scores indicate a higher likelihood of using the tool after the study is over.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Making Tool
Number analyzed (Participants) | 21
units on a scale | 3.43 (1.1)

7. Secondary Outcome: Feasibility - Ease of Use
Description: Ease of use refers to how easy an intervention is to use. In this study, we measures ease of use of the tool with a self-report, single item rated on Likert scales ranging from 1 (very hard) to 5 (very easy). A higher rating means the tool was considered easier to use.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Making Tool
Number analyzed (Participants) | 21
units on a scale | 4.4 (1.0)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: No more than minimal risk study.
Arm/Group | Decision Making Tool
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT04872569/Prot_SAP_000.pdf